CLINICAL TRIAL: NCT07052227
Title: The Influences of Blood Flow Restriction on Leg Press Perceptual Responses and Performance, and Systemic Arterial Stiffness
Brief Title: The Influences of Blood Flow Restriction on Leg Press
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Salisbury University (Other)
Responsible Party: Principal Investigator, Timothy Werner, Professor, Salisbury University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: #492
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Delfi Cuff; Fitcuff; Placebo - Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Delfi (Experimental)
  Interventions: Device: Delfi blood flow restriction cuff
- Fitcuff (Experimental)
  Interventions: Device: Fitcuffs
- Control (Placebo Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Device: Delfi blood flow restriction cuff — Leg press exercise with Delfi blood flow restriction cuff
  Arms: Delfi
Device: Fitcuffs — Leg press exercise with Fitcuff blood flow restriction cuff
  Arms: Fitcuff
Other: Control — Leg press exercise with no blood flow restriction cuff
  Arms: Control

SUMMARY:
This study will investigate the use of different blood flow restriction cuffs during leg press exercise on arterial stiffness, muscle morphology, performance, and participant perception.

DETAILED DESCRIPTION:
This study aims to investigate the use of Delfi vs. Fitcuffs blood flow restriction (BFR) cuff exercise on indices of arterial stiffness, muscle morphology, performance, and participant perception. Thirty adults aged 18-40 years old will undergo three treatment sessions (control (no BFR), Delfi BFR, and Fitcuffs BFR) in a randomized order separated by one week. A familiarization session will also occur one week before starting the treatment period. Each subject will undergo a series of tests including anthropometry, applanation tonometry, ultrasonography of the vastus lateralis, blood pressure acquisition, body composition, and maximal strength assessments (1RM). The exercise trial will consist of sets of leg press exercises performed to failure with a 2-second concentric and 2-second eccentric cadence at 20% of their 1RM using 60% of the supine limb occlusion pressure (LOP) with 1-minute rest intervals. Assessments will be performed immediately before and after the exercise bout during each treatment session. Two-way ANOVAs will be used to examine the main effects of treatment and treatment-order interaction on pulse wave velocity, muscle cross-sectional area, and perceptual response.

ELIGIBILITY:
Inclusion Criteria:

1. Physically active (> 1,000 MET/min/wk) for at least six months.
2. Weight stable for previous 6 months (+/-2.5 kg)

Exclusion Criteria:

1. Stage 2 hypertension (SBP >/= 140 and/or DBP >/= 90 mmHg)
2. BMI>40 kg/m2
3. Diabetes
4. Familial hypercholesterolemia
5. Past or current history of CHD, stroke or major CVD events. Respiratory diseases (not including asthma), endocrine or metabolic, neurological, or hematological disorders that would compromise the study or the health of the subject.
6. Participants must not be pregnant, plan to become pregnant during the study, or be nursing
7. Active renal or liver disease
8. All medications and supplements that influence dependent variables*
9. Recent surgery < 2 months
10. Alcohol abuse
11. Sleep apnea

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-14 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity | 10 minutes before and 10 minutes after the exercise intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Salisbury University, Salisbury, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Excel spreadsheet with data will be shared upon request.
Supporting Information: Study Protocol, SAP, Analytic Code